CLINICAL TRIAL: NCT04494815
Title: A Phase 1b, Randomised, Double-blind, Placebo- and Active Controlled, Single Dose Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of SR419 in Patients With Peripheral Neuropathic Pain
Brief Title: A Phase 1b Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of SR419
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai SIMR Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SR419-102
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2024-11

CONDITIONS: Peripheral Neuropathic Pain
Keywords: DPN, PHN...etc.

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treatment A (Experimental): Treatment A: Single 20 mg oral suspension dose of SR419 + single active control placebo capsule.
  Interventions: Drug: SR419; Drug: active control placebo
- Treatment B (Active Comparator): Treatment B: Single SR419 placebo oral suspension + single 300 mg oral capsule of active control.
  Interventions: Drug: active control; Drug: SR419 placebo
- Treatment C (Placebo Comparator): Treatment C: Single SR419 placebo oral suspension + single active control placebo capsule.
  Interventions: Drug: active control; Drug: active control placebo

INTERVENTIONS:
Drug: SR419 — Each participant will receive 1 dose of 20 mg SR419 oral suspension.
  Arms: Treatment A
Drug: active control — Each participant will receive 1 dose of 300 mg active control capsule.
  Arms: Treatment B; Treatment C
Drug: SR419 placebo — Each participant will receive 2 doses of SR419 placebo oral suspension.
  Arms: Treatment B
Drug: active control placebo — Each participant will receive 2 doses of active control placebo capsule.
  Arms: Treatment A; Treatment C

SUMMARY:
This study is to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of SR419 in Patients with Peripheral Neuropathic Pain

DETAILED DESCRIPTION:
This is a three-period, complete crossover, double-blind, randomised, placebo- and active-controlled study to compare the preliminary efficacy of a single dose of SR419 to placebo and active control in patients with peripheral neuropathic pain. The study also aims to evaluate the safety, tolerability, and PK of single doses of SR419 in patients with peripheral neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years at the time of informed consent.
2. Be diagnosed as suffering from chronic peripheral neuropathic pain, and specifically PHN or DPN.
3. Average daily pain over the last week prior to Screening to be of at least moderate severity (a score of ≥4 on the 11-point numeric rating scale [NRS]) and be of face, limb or torso location.
4. A minimum score of 19 on the pain DETECT questionnaire.

Exclusion Criteria:

1. Being pregnant or lactating at Screening or planning to become pregnant (self or partner) at any time during the study.
2. Prior or ongoing medical conditions, medical history, physical findings, or laboratory abnormality.
3. Known or suspected intolerance or hypersensitivity to any of the study drugs, close related compounds, or any of the stated ingredients.
4. Participants on controlled-release opioids (e.g., morphine) unless on a stable dose of Morphine Equivalent Dose (assessed by the Faculty of Pain Medicine Opioids Calculator) of up to and including 60 mg/day, at the discretion of the Investigator. Participants on instant-release opioids (e.g., codeine, oxycodone) must withhold dosing for 12 hours prior to administration of study drug.
5. Positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
6. Creatinine clearance as estimated by estimated glomerular filtration rate (eGFR) <60 mL/min.
7. A history of major psychiatric disorder(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
QST of an affected area. | Up to Day18(-2~+5) for the safety follow up since Day1
  QST: Quantitative sensory testing

SECONDARY OUTCOMES:
The incidence, frequency, and severity of TEAEs. | Up to Day18(-2~+5) for the safety follow up since Day1
  TEAE: Treatment-Emergent Adverse Events
Spontaneous pain score | Up to Day18(-2~+5) for the safety follow up since Day1
  Pain score will be assessed via painDETECT questionnaire with a value range of 0~38, which includes three situations: If a subject gets a score of 0~12, it means a neuropathic pain component is unlikely(less than 15% probability); if a score of 13~19, it means the result is ambiguous, however, a neuropathic pain component can be present; if the score is equal to or greater than nineteen, it means a neuropathic pain is likely(more than 90% probability).
QST of an unaffected area. | Up to Day18(-2~+5) for the safety follow up since Day1
Plasma concentration of SR419 after dosing. | Up to Day11(+3)

CONTACTS AND LOCATIONS:
Overall Officials: Kai Wu, Study Director — SIMR
Locations (1):
- Clinical Research Facility Medical School, University of Adelaide, Adelaide, South Australia, Australia